CLINICAL TRIAL: NCT04964037
Title: Analysis of Relationship Between Metabolic Biomarkers and Efficacy of Systemic Glucocorticoid in Acute Exacerbation of COPD
Brief Title: Analysis of Relationship Between Metabolic Biomarkers and Efficacy of Glucocorticoid in AECOPD
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Liang Ying, Peking University Third Hospital, Peking University Third Hospital
Other Study IDs: LM2018024
Record Dates: First submitted 2021-06-29; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum sample was obtained before glucocorticoid was given to the subject.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment success group: No intervention
  Interventions: Other: No intervention
- Treatment failure group: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Evidences have shown that systemic glucocorticoid cannot not be benefit to all of the patients with AECOPD. The problem that how the clinicians can screen the patients who can benefit from systemic glucocorticoid needs to be solved. Our previous study found that serum metabolites profile in COPD patients differed from that in controls. Therefore, we hypothesized that metabolome changes in patients with AECOPD may be associated with the efficacy of systemic glucocorticoid. In this study, we will utilize ultraperformance liquid chromatography / mass spectrometry (LC-MS) and gas chromatography / mass spectrometry (GC-MS) methods for analysis of the metabolites in AECOPD patients and compare the metabolites profiles between patients with systemic glucocorticoid treatment success and treatment failure. We aim to detect the metabolic biomarkers and metabolic pathways which are related to efficacy of systemic glucocorticoid and contribute to the precise treatment of COPD.

DETAILED DESCRIPTION:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) significantly increases the mortality of the patients with COPD. Guidelines have recommended systemic glucocorticoid as regular treatment. Recently, evidences have shown that systemic glucocorticoid cannot not be benefit to all of the patients with AECOPD. Thus the problem that how the clinicians can screen the patients who can benefit from systemic glucocorticoid needs to be solved urgently. A previous study found that plasma metabolome changed significantly after dexamethasone treatment in health participants. Furthermore, inter-person variability was high and remained uninfluenced by treatment, suggesting the potential of metabolomics for predicting the efficacy and side effects of systemic glucocorticoid. Our previous study found that serum metabolites profile in COPD patients differed from that in controls. Therefore, we hypothesized that metabolome changes in patients with AECOPD may be associated with the efficacy of systemic glucocorticoid. In this study, we will utilize ultraperformance liquid chromatography / mass spectrometry (LC-MS) and gas chromatography / mass spectrometry (GC-MS) methods for analysis of the metabolites in AECOPD patients and compare the metabolites profiles between patients with systemic glucocorticoid treatment success and treatment failure. We aim to detect the metabolic biomarkers and metabolic pathways which are related to efficacy of systemic glucocorticoid and contribute to the precise treatment of COPD.

ELIGIBILITY:
Inclusion Criteria:

* All the patients met the diagnosis of COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines and had definite airflow limitation with a post-bronchodilator forced expiratory volume in 1 second (FEV1) / forced vital capacity (FVC)<0.7.
* They were admitted to the ward of Department of Respiratory and Critical Care Medicine due to COPD exacerbation.

Exclusion Criteria:

* age <40 years;
* subjects with airway diseases other than COPD;
* comunity acquired pneumonia;
* active tuberculosis;
* severe liver or renal dysfunction;
* malignancy;
* HIV infection or immunodeficiency;
* ever received glucocorticoid in the past month.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively recruited the patients admitted to the ward of Department of Respiratory and Critical Care Medicine due to COPD exacerbation from January 2017 to March 2018
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Serum metabolic biomarkers | Through study completion, an average of 10 days
  Liquid chromatography / mass spectrometry (LC-MS) was used to analyze the metabolites in AECOPD patients.